CLINICAL TRIAL: NCT02529709
Title: The Effect of Meal Composition on Blood Lipid Concentrations
Brief Title: The Effect of Meal Composition on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Meena Shah, Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TexasCU
Record Dates: First submitted 2015-08-14; First posted 2015-08-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-protein meal condition (Experimental)
  Interventions: Other: High-Protein Condition
- High-monounsaturated fat meal condition (Active Comparator)
  Interventions: Other: High-Monounsaturated Fat Condition

INTERVENTIONS:
Other: High-Protein Condition — The participants will be fed a high-protein meal
  Arms: High-protein meal condition
Other: High-Monounsaturated Fat Condition — The participants will be fed a high-monounsaturated fat meal
  Arms: High-monounsaturated fat meal condition

SUMMARY:
The purpose of this study is to see if a high-protein meal leads to a better postprandial (after a meal) blood lipid profile compared to a high-monounsaturated meal.

DETAILED DESCRIPTION:
The effect of a high-protein diet compared to a high-monounsaturated fat diet on fasting lipids is controversial (1,2), In addition, these studies did not examine the effect of a high-protein compared to a high-monounsaturated meal on postprandial lipid concentrations. Postprandial lipid responses are important to examine since they are associated with heart disease (3,4). In addition, most individuals in Western countries are in a postprandial state for majority of the day. The present study will compare the effect of a high-protein meal versus a high-monounsaturated fat meal on postprandial lipid responses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-65 years.

Exclusion Criteria:

* Use of medications or supplements that affect lipid levels, body weight, or blood glucose,
* following a weight loss diet,
* being a vegan,
* smoking,
* heavy alcohol use,
* pregnancy,
* lactation,
* severe depression,
* eating disorders,
* presence of liver, kidney, gastrointestinal, adrenal, or untreated thyroid disease,
* diabetes,
* lactose intolerance,
* documented mal-absorption, or
* bowel surgery that affects absorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Blood lipid concentrations. | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins

SECONDARY OUTCOMES:
IL-6 | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
TNF-α | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
C-reactive protein | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
GLP-1 | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
Insulin | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
Glucagon | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
Glucose | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins
Leptin | At 0 minute before the meal begins and at 30, 60, 120, and 180 minutes after the meal begins

CONTACTS AND LOCATIONS:
Overall Officials: Meena Shah, Ph.D., Principal Investigator — Tzu Chi University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

REFERENCES:
- [Background] Appel LJ, Sacks FM, Carey VJ, Obarzanek E, Swain JF, Miller ER 3rd, Conlin PR, Erlinger TP, Rosner BA, Laranjo NM, Charleston J, McCarron P, Bishop LM; OmniHeart Collaborative Research Group. Effects of protein, monounsaturated fat, and carbohydrate intake on blood pressure and serum lipids: results of the OmniHeart randomized trial. JAMA. 2005 Nov 16;294(19):2455-64. doi: 10.1001/jama.294.19.2455. PMID 16287956
- [Background] Luscombe-Marsh ND, Noakes M, Wittert GA, Keogh JB, Foster P, Clifton PM. Carbohydrate-restricted diets high in either monounsaturated fat or protein are equally effective at promoting fat loss and improving blood lipids. Am J Clin Nutr. 2005 Apr;81(4):762-72. doi: 10.1093/ajcn/81.4.762. PMID 15817850
- [Background] Simons LA, Dwyer T, Simons J, Bernstein L, Mock P, Poonia NS, Balasubramaniam S, Baron D, Branson J, Morgan J, et al. Chylomicrons and chylomicron remnants in coronary artery disease: a case-control study. Atherosclerosis. 1987 May;65(1-2):181-9. doi: 10.1016/0021-9150(87)90020-7. PMID 3496893
- [Background] Bansal S, Buring JE, Rifai N, Mora S, Sacks FM, Ridker PM. Fasting compared with nonfasting triglycerides and risk of cardiovascular events in women. JAMA. 2007 Jul 18;298(3):309-16. doi: 10.1001/jama.298.3.309. PMID 17635891